CLINICAL TRIAL: NCT01060696
Title: Efficacy of Mefenamic Acid and Hyoscine for Pain Relief During Saline Infusion Sonohysterography in Infertile Women. A Double Blind Randomized Controlled Trial
Brief Title: Efficacy of Mefenamic Acid and Hyoscine for Pain Relief During Saline Infusion Sonohysterography in Infertile Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Singpetch Suksompong, Mahidol University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 615/2551
Record Dates: First submitted 2010-01-31; First posted 2010-02-02 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Infertility
Keywords: Infertility; Saline infusion sonohysterography; Pain; Hyoscine; Mefenamic acid; women
MeSH Terms: conditions — Infertility; Pain | interventions — Mefenamic Acid; Scopolamine; Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyoscine, Mefenamic acid, Placebo (Experimental): Blind randomization to three groups. Mefenamic acid group Hyoscine group Placebo group
  Interventions: Drug: Mefenamic acid or Hyoscine or placebo

INTERVENTIONS:
Drug: Mefenamic acid or Hyoscine or placebo — Mefenamic acid 500 mg. single oral use 30 minutes before SIS Hyoscine 10 mg. single oral use 30 minutes before SIS Placebo single oral use 30 minutes before SIS
  Other Names: Ponstan (Mefenamic acid); Buscopan (Hyoscine-N-butylbromide)

SUMMARY:
The infertility patients who are performed saline infusion sonohysterography (SIS) for studying the pathology inside the uterine cavity has pain. From pilot study the pain score is 6.80. It will have more benefits if we can manage this procedure with less or no pain. Many studies have tried to decrease pain such as types of catheter, intrauterine lidocaine infusion. Some have real effects but no study with oral Mefenamic acid or Hyoscine before the procedure.The drugs are safe and easy to administration and chief.

ELIGIBILITY:
Inclusion Criteria:

* infertility female
* no history of HSG or Hysteroscopy

Exclusion Criteria:

* vaginal or pelvic infection
* abnormal Pap smear
* contraindications for Mefenamic acid including upper and lower GI ulcers, bleeding disorder, Asthma or allergies, renal disease, using Warfarin,Aspirin, Lithium, history of Mefenamic acid or Hyoscine allergies

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-03 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Pain relief by oral Mefenamic acid or Hyoscine and placebo during saline infusion sonohysterography | Before, during and after the procedure

SECONDARY OUTCOMES:
Patients satisfaction during saline infusion sonohysterography | After the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Singpetch Suksompong, Doctor, Principal Investigator
Locations (1):
- Siriraj hospital Mahidol university, Bangkok, Bangkok, Thailand